CLINICAL TRIAL: NCT01845623
Title: A Randomized, Double-blind, Double-dummy, Placebo-controlled, 3-period Crossover Study to Evaluate the Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of Orally Inhaled Indacaterol Administered Via the EPIC Test Fixture and the Concept1 Device in Adult Patients With Persistent Asthma
Brief Title: A Study to Evaluate the Effects of Indacaterol Maleate (QAB149) as a New Formulation in the EPIC Test Fixture
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CMID001A2201; 2011-001824-39 (EudraCT Number)
Record Dates: First submitted 2013-04-17; First posted 2013-05-03 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2013-07

CONDITIONS: Asthma
Keywords: Asthma; Indacaterol; QAB149
MeSH Terms: conditions — Asthma | interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Experimental)
  Interventions: Drug: QAB149 75 mg Concept 1; Other: Placebo EPIC Test Fixture
- Treatment B (Experimental)
  Interventions: Drug: QAB149 75 mg Epic Test Fixture; Other: Placebo Concept 1
- Treatment C (Placebo Comparator)
  Interventions: Other: Placebo Concept 1; Other: Placebo EPIC Test Fixture

INTERVENTIONS:
Drug: QAB149 75 mg Concept 1 — QAB149 delivered via the concept 1 device.
  Arms: Treatment A
Drug: QAB149 75 mg Epic Test Fixture — QAB149 delivered via the EPIC test fixture
  Arms: Treatment B
Other: Placebo Concept 1 — Placebo administered via the Concept 1 device.
  Arms: Treatment B; Treatment C
Other: Placebo EPIC Test Fixture — Placebo administered via the EPIC Test Fixture.
  Arms: Treatment A; Treatment C

SUMMARY:
This study will assess the pharmacodynamics, safety, tolerability and pharmacokinetics of indacaterol maleate (QAB149), administered via the EPIC test fixture. The study aims to determine whether the novel device has a similar clinical profile as the established concept 1 device.

ELIGIBILITY:
Inclusion Criteria:

Male and female patients with asthma, aged 18 or above Patients using inhaled corticosteroid (with or without long acting beta agonist) Patients who demonstrate an increase in FEV1 after inhaling a short acting beta agonist

Exclusion Criteria:

Asthma exacerbations in previous 6 months COPD or other pulmonary disease Excessive use of short acting beta agonists

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Trough Forced Expiratory Volume in 1 Second (FEV1) Following 3 Days of Treatment | Day 4
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 was defined as the mean of two measurements at 23h 10min and 23h 45min post the Day 3 dose.

SECONDARY OUTCOMES:
Peak Forced Expiratory Volume in 1 Second (FEV1) on Days 1 and 3 | Days 1 and 3
  Spirometry was conducted according to internationally accepted standards. Peak FEV1 is the maximum FEV1 recorded in the period between 5 minutes and 4 hours post dose on Days 1 and 3.
Time to Peak Forced Expiratory Volume in 1 Second (FEV1) on Days 1 and 3 | Days 1 and 3
  Spirometry was conducted according to internationally accepted standards. Peak FEV1 is the maximum FEV1 recorded in the period between 5 minutes and 4 hours post dose on Days 1 and 3.
Forced Vital Capacity (FVC) at Each Time-point on Day 1, 2, 3 and 4 | Days 1, 2, 3 and 4
  Spirometry was conducted according to internationally accepted standards. FVC was calculated at each time point up to 4 hours post-dose and at 23 hours 10 min and 23 hours 45 min on Days 1/2 and 3/4.
Forced Expiratory Volume in 1 Second (FEV1) Standardized (With Respect to Length of Time) Area Under the Curve (AUC) From pre-dose to 4 hours post dose on Days 1 and 3 | Days 1 and 3
  FEV1 was measured with spirometry conducted according to internationally accepted standards. Measurements were made at 5, 15, and 30 minutes; and 1, 2, 3 and 4 hours post-dose. The standardized AUC FEV1 was calculated as the sum of trapezoids divided by the length of time.
Peak Expiratory Flow Rate measured daily each morning and evening. | Morning and evening from screening to study completion (up to 86 days)
  Peak Expiratory Flow (PEF) was measured every morning and evening from screening until study completion using a peak flow meter, and was recorded in the patient diary.
Forced Expiratory Volume in 1 Second (FEV1) | Days 1, 2, 3 and 4
  Spirometry was conducted according to internationally accepted standards. Forced expiratory volume in 1 second (FEV1) is the amount of air that can be exhaled in one second. FEV1 was measured at each time point up to 4 hours on Days 1 and 3 and at 23hours 10 mins and 23 hours 45 mins on Days 2 and 4.
Ratio of Forced Expiratory Volume in 1 Second (FEV1) and Forced Vital Capacity (FVC) (FEV1/FVC | Days 1, 2, 3, 4
  Spirometry was conducted according to internationally accepted standards. FEV1/FVC represents the proportion of the total amount of air that is exhaled from the lungs during the first second of forced exhalation. FEV1/FVC was measured at each timepoint up to 4 hours on Days 1 and 3 and 23hours 10mins and 23hours 45 mins on Days 2 and 4.
Forced expiratory Flow 25-75% (FEF25-75%) | Days 1, 2, 3, 4
  The forced expiratory flow (FEF) 25%-75% measurement describes the amount of air expelled from the lungs during the middle half (25% - 75%) of the forced vital capacity test and is measured using spirometry. FEF 25-75% was measured at each timepoint up to 4 hours on Days 1 and 3 and 23hours 10mins and 23hours 45 mins on Days 2 and 4
Number of puffs of rescue medication used | Everyday from screening to study completion (up to 86 days)
  Participants maintained a diary to record the daily number of puffs of rescue Short-acting B2 agonist (SABA) used to treat asthma symptoms.
The number of participants with adverse events used as a measure of Safety and Tolerability | Baseline to study completion (up to 59 days)
  Safety and tolerability of indacaterol administered via the EPIC test fixture and the Concept1 was measured by collecting the following safety data: - number and percentage of adverse events reported by participants for the duration of the study - safety laboratory testing - measurement of vital signs (blood pressure and heart rate) - measurement of ECGs
AUC (0-24) - area under the serum concentration-time curve | Day 1 and Day 3 (pre-dose, 5, 15, 30 mins, 1, 2, 4, 8, 12, 24hours post dose
  The PK parameter AUC0-24 - area under the serum concentration-time curve - was determined from the serum concentration time profile of indacaterol on Days 1 and 3 from time zero to 24 hours post dose using a non-compartmental method
Cmax - observed maximum serum concentration following drug administration | Day 1 and Day 3 (pre-dose, 5, 15, 30 mins, 1, 2, 4, 8, 12, 24hours post dose
  The PK parameter Cmax - observed maximum serum concentration following drug administration - was determined from the serum concentration time profile of indacaterol on Days 1 and 3 using a non-compartmental method.
Tmax - time to reach maximum concentration after drug administration | Day 1 and Day 3 (pre-dose, 5, 15, 30 mins, 1, 2, 4, 8, 12, 24hours post dose
  The PK parameter Tmax - time to reach maximum concentration after drug administration - was determined from the serum concentration time profile of indacaterol on Days 1 and 3 using a non-compartmental method.
Racc - accumulation ratio of exposure (AUC0-24 and Cmax) on Day 3 relative to Day 1 | Day 1 and Day 3 (pre-dose, 5, 15, 30 mins, 1, 2, 4, 8, 12, 24hours post dose
  The PK parameter Racc - accumulation ratio of exposure (AUC0-24 and Cmax) on Day 3 relative to Day 1 - was determined from the serum concentration time profile of indacaterol on Days 1 and 3 using a non-compartmental method.
Trough Forced Expiratory Volume in 1 Second (FEV1) Following 1 Day of Treatment | Day 2
  FEV1 is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing. The trough in FEV1 was defined as the mean of two measurements at 23h 10min and 23h 45min post the Day 1 dose.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals